CLINICAL TRIAL: NCT07110506
Title: Comparison of Hemodynamic Variables Between Using Conventional Invasive Catheter Monitoring and Non-invasive Piezoelectric Sensor
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 202459
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Monitoring

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invasive group (Active Comparator): Arterial pressure is obtained from invasive arterial monitoring
  Interventions: Other: Arterial pressure monitoring
- Noninvasive arterial monitoring (Experimental): Arterial pressure is obtained from non-invasive arterial monitoring
  Interventions: Other: Arterial pressure monitoring

INTERVENTIONS:
Other: Arterial pressure monitoring — Arterial pressure is monitored and obtained

SUMMARY:
Arterial pressure is obtained from invasive arterial monitoring and noninvasive arterial monitoring using piezoelectric sensor and compared.

ELIGIBILITY:
Inclusion Criteria:

* Cases who require Invasive arterial pressure monitoring d/t bleeding.

Exclusion Criteria:

* Patients with cardiovascular disease, cerebrovascular diseases, renal disease, or Marfan syndrome
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2026-12-18 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Arterial pressure | For 30 min after the induction of anesthesia,
  After the induction of anesthesia, 20G catheter is placed for invasive arterial pressure monitoring in the radial artery and pressure sensor is attached for noninvasive arterial pressure monitoring in the contralateral radial artery. Then, invasive and noninvasive arterial pressures are monitored and obtained simultaneously.

IPD SHARING:
Plan to Share IPD: No